CLINICAL TRIAL: NCT03741335
Title: Group Exercise Training for Fall Prevention and Functional Improvements During and After Treatment for Prostate Cancer
Brief Title: GET FIT Prostate: A Randomized Controlled Exercise Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00018354; NCI-2019-01422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018354 (Other: OHSU Knight Cancer Institute); R01CA222605 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-14 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Resistance Training; Tai Ji

STUDY DESIGN:
Intervention Model Description: 3-group, single-blind, parallel design randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the participants assigned study arm. Participants will not be formally masked from knowing whether or not they are assigned to an experimental or control group, but every effort will be made not to overemphasize expected outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength Training (Experimental): Participants wear a weighted vest while performing exercises using functional movement patterns used in everyday activities (chair rises, 90° squats, side-to-side squats, toe raises, lunges (forward, lateral, backward, walking), multi-directional step ups). Participants attend supervised, group-based moderate-intensity strength training program remotely 3 times per week for 60 minutes per session.
  Interventions: Other: Resistance Training
- Stretching Control (Active Comparator): Participants attend a supervised flexibility program where they will perform a series of whole body stretching exercises with a focus on developing and maintaining a healthy back. Participants attend a supervised, group-based supervised flexibility program remotely 3 times per week for 60 minutes per session.
  Interventions: Other: Stretching
- Tai Ji Quan Training (Experimental): An integrated exercise routine consisting of 8 purposeful movement forms and a set of therapeutic movements. Participants attend a supervised, group-based tai ji quan program remotely where they perform an integrated exercise routine consisting of 8 purposeful movement forms and a set of therapeutic movements 3 times per week for 60 minutes per session.
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Resistance Training — Participants attend supervised, group-based moderate-intensity strength training program 3 times per week for 60 minutes per session.
  Other Names: Strength Training
  Arms: Strength Training
Other: Stretching — Participants attend a supervised, group-based supervised flexibility program 3 times per week for 60 minutes per session
  Arms: Stretching Control
Other: Tai Chi — Participants attend a supervised, group-based tai ji quan program where they perform an integrated exercise routine consisting of 8 purposeful movement forms and a set of therapeutic movements 3 times per week for 60 minutes per session.
  Arms: Tai Ji Quan Training

SUMMARY:
The GET FIT Prostate trial (Group Exercise Training for Fall prevention and functional Improvements during and after Treatment for Prostate cancer) is a single-blind, parallel group, randomized controlled trial comparing - 1) tai ji quan (functional balance) and 2) strength training (functional strength) against each other and vs. 3) a stretching control (functional mobility) - over a 6-mos. supervised intervention and 6-mos. follow-up. Two million prostate cancer survivors are alive in the U.S. and nearly half (45%) will receive androgen deprivation therapy (ADT) to reduce tumor androgen exposure and slow down cancer progression. While beneficial for cancer survival, significant treatment-induced side effects from ADT may lead to serious health consequences including falls, frailty, and dysfunction that contribute to morbidity and mortality

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine and compare the efficacy of tai ji quan training and strength training in reducing the incidence of falls in prostate cancer survivors on antiandrogen therapy (ADT).

SECONDARY OBJECTIVE:

I. To determine and compare the efficacy of tai ji quan training and strength training to reduce frailty and dysfunction in prostate cancer survivors on ADT.

TERTIARY OBJECTIVE:

I. To determine how well the benefits of tai ji quan and strength interventions persist over a 6-month period.

EXPLORATORY OBJECTIVE:

I. To explore the patterns and predictors of types of men (including host and treatment factors) who benefit most from tai ji quan and strength training.

OUTLINE:

The study is a 3-group, single-blind, parallel design randomized controlled trial in prostate cancer survivors treated with ADT. Participants in each study group will attend supervised 1-hr classes, 3 days a week for 6 months.

ARM 1: Tai ji quan, an integrated exercise routine consisting of 8 purposeful movement forms and a set of therapeutic movements, specifically designed to challenge limits of stability and train gait patterns, as reflected in movements such as upright trunk positioning, displacement of body's center of mass over the weight-bearing leg, and step initiation, locomotion, and termination.

ARM 2: Strength training. Participants wear a weighted vest while performing exercises using functional movement patterns that challenge balance by using muscle groups and movement involved in everyday activities (chair rises, 90°squats, side-to-side squats, toe raises, lunges (forward, lateral, backward, walking), multi-directional step ups).

ARM 3: Stretching control. Participants in the control group will attend a supervised flexibility program of the same total weekly duration as the experimental arms (e.g., 3, 60-min sessions per week). Control participants will perform a series of whole body stretching exercises, according to the ACSM guidelines for flexibility training, with a focus on developing and maintaining a healthy back.

Six Month Follow-Up: Participants will be followed for an additional 6 months after the 6-month supervised intervention stops to track falls (using same monthly report used during intervention phase). Exercise questionnaires to track participation in home or community exercise programs and will be collected at the 9- and 12-month time periods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically confirmed prostate cancer (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his physician.)
* Currently on ADT for >= 6 months OR not currently receiving ADT, but received >= 6-month course within the last 10 years (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his physician.)
* If they have had other treatment, such as surgery, radiation or chemotherapy, it must have been completed >= 6 weeks prior to enrollment and no concurrent adjuvant therapy other than ADT for prostate cancer (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his physician).
* Meets criteria for having experienced >= 1 fall in the last year (confirmed by self-report on Health History Questionnaire) or if no falls, meets criteria for slow Timed Up and Go (TUG) time (>= 12.0 seconds) OR slow chair stand time (>= 10.0 seconds) (confirmed by baseline screening testing).

Exclusion Criteria:

* Current participation in moderate or vigorous lower-body strength training two or more times per week for 30 minutes or more or participating in tai chi two or more times per week for 30 minutes or more (confirmed by self-report on Health History Questionnaire or by discretion of the principal investigator).
* Cognitive difficulties that preclude answering the survey questions, participating in the exercise classes or performance tests, or providing informed consent (Confirmed by the professional opinion of the principal investigator, Dr. Kerri Winters-Stone.).
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in moderate intensity exercise (Confirmed by self-report on the Health History Questionnaire, and/or by physician clearance. If in the professional opinion of the principal investigator, Dr. Kerri Winters-Stone, contraindications other than those identified by the patient or physician are present, she may consider the participant ineligible.).
* Not medically cleared for participation in moderate intensity exercise. (Confirmed by physician clearance.).
* Knowingly unable to attend > 75% of the intervention classes due to conflict with the designated time of day, days of the week, and/or location for the exercise class which they initially enrolled. (Confirmed by documentation in the Case Report Form titled "CRF - Participant Contact Info_GET FIT Prostate").
* Not fluent in English and therefore incapable of answering survey questions, participating in class, following directions during performance testing, and providing informed consent when English is the language used. (Confirmed by documentation in the Case Report Form titled "CRF - Participant Contact Info_GET FIT Prostate" or the professional opinion of the principal investigator, Dr. Kerri Winters-Stone.).

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual quantitative participant data collected during the trial, after deidentification.
Time Frame: Beginning 3 months following final publication
Access Criteria: Access will be provided to investigators who provide a methodologically sound proposal and complete a data sharing agreement that includes commitments to: (1) using the data only for research purposes and not to identify any individual participant, (2) securing the data using appropriate computer technology, and (3) destroying or returning the data after analyses are completed.
  Proposals should be directed to wintersk@ohsu.edu. To gain access to data, data requestors will need to sign a data sharing agreement.

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Winters-Stone KM, Li F, Horak F, Dieckmann N, Hung A, Amling C, Beer TM. Protocol for GET FIT Prostate: a randomized, controlled trial of group exercise training for fall prevention and functional improvements during and after treatment for prostate cancer. Trials. 2021 Nov 6;22(1):775. doi: 10.1186/s13063-021-05687-7. PMID 34742325
- [Derived] Winters-Stone KM, Boisvert C, Li F, Lyons KS, Beer TM, Mitri Z, Meyers G, Eckstrom E, Campbell KL. Delivering exercise medicine to cancer survivors: has COVID-19 shifted the landscape for how and who can be reached with supervised group exercise? Support Care Cancer. 2022 Mar;30(3):1903-1906. doi: 10.1007/s00520-021-06669-w. Epub 2021 Nov 6. PMID 34741653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-dwelling prostate cancer survivors were recruited between February 2019 and September 2022. The first participant was enrolled on the 5th of February 2019 and the last participant was enrolled on the 19th of September 2022.
Pre-assignment Details: 284 men met eligibility criteria and were randomized to receive one of three treatment arms as specified per protocol.
Period: Overall Study
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Started | 97 | 92 | 95
Completed | 82 | 73 | 72
Not Completed | 15 | 19 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training | Total
Number analyzed (Participants) | 97 | 92 | 95 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (6.7) | 72.4 (7.4) | 73.0 (7.1) | 72.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 97 | 92 | 95 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 6
  Not Hispanic or Latino | 95 | 84 | 90 | 269
  Unknown or Not Reported | 2 | 5 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 7
  White | 90 | 84 | 85 | 259
  More than one race | 2 | 2 | 3 | 7
  Unknown or Not Reported | 3 | 3 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 97 | 92 | 95 | 284

OUTCOME MEASURES:

1. Primary Outcome: Number of Falls
Description: Prospective assessment of falls will be done by collecting monthly reports returned by postal and/or electronic mail. A fall is defined as unintentionally coming to rest on the ground or at some other lower level, not as a result of a major intrinsic event (e.g., stroke or syncope) or overwhelming hazard.
Time Frame: Baseline up to 6 months
Measure: Mean (95% Confidence Interval); unit: Average fall count per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 94 | 84 | 85
Average fall count per 6 months | 0.29 [.18 to .47] | .33 [.21 to .54] | .38 [.24 to .60]

2. Secondary Outcome: Change in Total Frailty Score
Description: Frailty will be measured using the components of the Frailty Phenotype, which consist of measures of lean body mass, fatigue, physical activity, walk speed, and muscle strength, listed as additional outcomes below. Each component of frailty is assessed using measures that will capture frailty criteria in the prostate cancer survivor population using appropriate cutoff scores indicating that a component meets a particular criterion. A total frailty score was calculated for each patient at each timepoint defined as a count of the number of frailty components met.
Time Frame: Baseline up to 12 months
Measure: Number (95% Confidence Interval); unit: Incidence rate ratio
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 84 | 77 | 80
Incidence rate ratio
  Baseline-6mo | .41 [.06 to .76] | .84 [.56 to 1.20] | .66 [.36 to .97]
  6mo-12mo | 1.66 [1.28 to 2.04] | .99 [.69 to 1.31] | 1.16 [.83 to 1.49]

3. Secondary Outcome: Lean Body Mass
Description: Lean body mass will be measured by bioelectric impedance analysis (in kg). Higher values indicate higher lean body mass.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 75 | 63 | 66
Score on a scale per 6 months
  Baseline-6mo | -.03 [-.72 to .66] | -.68 [-1.42 to .07] | -.87 [-1.64 to -.10]
  6mo-12mo | -.18 [-1.15 to .79] | -.34 [-1.43 to .75] | -.06 [-1.11 to .99]

4. Secondary Outcome: Fatigue-general
Description: Fatigue will be measured using the Short Form (SF)-36 Vitality scale. The scale ranges from 0-100 with lower scores indicating higher fatigue (i.e., less vitality).
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 97 | 91 | 94
Score on a scale per 6 months
  Baseline-6mo | 1.60 [.08 to 3.12] | -.63 [-2.21 to .95] | 1.47 [-.14 to 3.08]
  6mo-12mo | -1.26 [-2.56 to .04] | -.08 [-1.47 to 1.32] | .32 [-1.06 to 1.71]

5. Secondary Outcome: Fatigue-cancer
Description: Fatigue will also be measured using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). The questionnaire includes 13 items rated from "not at all" to "very much" over the past 7 days, and possible scores from 0 to 52. Lower scores indicate more fatigue, while higher scores indicate less severe fatigue.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 97 | 91 | 94
Score on a scale per 6 months
  Baseline-6mo | 1.79 [.54 to 3.05] | .51 [-.79 to 1.81] | 1.74 [.42 to 3.07]
  6mo-12mo | -1.15 [-2.51 to .20] | -.32 [-1.76 to 1.12] | .17 [-1.28 to 1.61]

6. Secondary Outcome: Physical Activity
Description: Physical activity will be measured by physical activity-related energy expenditure (kcals/week) calculated from self-report moderate-to-vigorous physical activity (MVPA). Lower scores indicate less MVPA and higher scores indicate more MVPA.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 97 | 91 | 94
Score on a scale per 6 months
  Baseline-6mo | 514.72 [-26.22 to 1055.67] | -702.11 [-1261.49 to -142.74] | -319.98 [-885.25 to 245.30]
  6mo-12mo | -710.9 [-1226.03 to -195.76] | 259.06 [-285.54 to 803.67] | 196.81 [-354.30 to 747.93]

7. Secondary Outcome: Walk Speed
Description: Walk speed will be measured by the 3-meter Timed Up and Go, a widely used clinical measure of functional mobility that evaluates the time it takes to rise from a chair, walk 3m, turn around, and return and sit in the chair.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 84 | 78 | 81
Score on a scale per 6 months
  Baseline-6mo | .11 [.08 to .15] | .07 [.04 to .11] | .09 [.06 to .13]
  6mo-12mo | -.03 [-.06 to 0.00] | -.02 [-.06 to .01] | -.02 [-.05 to .01]

8. Secondary Outcome: Muscle Strength
Description: Muscle strength will be measured by timed chair stand test (seconds required to rise from chair 5 times). The larger the time, the longer it took them to complete 5 chair stands.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 84 | 77 | 80
Score on a scale per 6 months
  Baseline-6mo | -2.63 [-3.45 to -1.81] | -2.15 [-3.00 to -1.28] | -1.85 [-2.73 to -.96]
  6mo-12mo | .76 [-.07 to 1.60] | 0.18 [-.72 to 1.08] | .75 [-.14 to 1.64]

9. Secondary Outcome: Change in Functional Mobility
Description: Functional mobility will be measured by the Timed Up and Go (TUG) test which measures the time that it takes a person to rise from a chair, walk 7 meters (m), turn around a cone and return and sit in the chair. Larger times means they were slower, and shorter times mean they were faster.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 84 | 78 | 80
Score on a scale per 6 months
  Baseline-6mo | -1.45 [-1.90 to -1.00] | -.61 [-1.08 to -.15] | -.93 [-1.40 to -.45]
  6mo-12mo | .60 [.20 to 1.00] | .14 [-.28 to .56] | .17 [-.24 to .59]

10. Secondary Outcome: Change in Functional Balance
Description: Functional balance will be measured by postural sway which evaluates how well a person can maintain their equilibrium during quiet standing. Participants will perform a standard 30-second postural sway test to measure the velocity (meters per second [m/s]) of sway during quiet standing with feet together and eyes closed using lightweight, inertial wireless sensors worn on the trunk. Lower sway velocity (m/s) indicates better postural stability.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 84 | 78 | 81
Score on a scale per 6 months
  Baseline-6mo | 0.00 [-.04 to .04] | .01 [-.04 to .05] | -.02 [-.06 to .03]
  6mo-12mo | -.02 [-.03 to .06] | .01 [-.03 to .06] | .02 [-.02 to .07]

11. Secondary Outcome: Change in Perceived Physical Function
Description: Perceived physical function will be measured by self-report using the physical function subscale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30; version 3, App. I). Scores on the subscale range from 0-100 where higher scores indicate better physical functioning.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 97 | 91 | 92
Score on a scale per 6 months
  Baseline-6mo | -1.02 [-3.50 to 1.45] | -.35 [-2.93 to 2.22] | -2.18 [-4.82 to .46]
  6mo-12mo | -1.27 [-3.95 to 1.41] | -.32 [-3.16 to 2.53] | 1.85 [-1.01 to 4.71]

12. Secondary Outcome: Flexibility
Description: Flexibility will be measured using the chair sit and reach. While seated on the edge of a chair, participants bend from the hip and reach toward or past the toes. The toes represent 0, so a reach short of the toes is recorded in negative inches, and a reach past the toes is recorded in positive inches. Higher negative values indicate greater flexibility.
Time Frame: Baseline up to 12 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
Number analyzed (Participants) | 85 | 80 | 84
Score on a scale per 6 months
  Baseline-6mo | 1.70 [.69 to 2.70] | 1.93 [.87 to 2.99] | 1.73 [.65 to 2.81]
  6mo-12mo | -1.11 [-1.88 to -.33] | -1.96 [-2.79 to -1.12] | -1.59 [-2.40 to -.77]

ADVERSE EVENTS:
Time Frame: Up to 1 year.
Description: An Adverse Event survey was created by the study team to be administered monthly during the participants' year-long participation in the study.
Arm/Group | Strength Training | Stretching Control | Tai Ji Quan Training
All-Cause Mortality (participants affected / at risk) | 2/97 | 4/92 | 1/95
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/92 | 3/95
Other Adverse Events (participants affected / at risk) | 0/97 | 0/92 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength Training (N=97) | Stretching Control (N=92) | Tai Ji Quan Training (N=95)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
New immunotherapy treatment (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03741335/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03741335/ICF_002.pdf